CLINICAL TRIAL: NCT00580229
Title: A Safety Analysis of Oral Prednisone as a Pre-Treatment for Rituximab in Rheumatoid Arthritis.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U4164s
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituxan; Rituximab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prednisone (Experimental): Prednisone 40mg by mouth 30-60 minutes prior to rituximab.
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: prednisone — prednisone 40mg by mouth 30-60 minutes prior to rituximab
  Other Names: Rayos

SUMMARY:
This study will be an open-label prospective analysis of oral prednisone (compared to IV methylprednisolone) as a pre-treatment for rituximab in patients with rheumatoid arthritis. The study will be useful as pilot data to establish that there are no different trends between the two treatment strategies at decreasing the frequency and severity of acute infusion reactions. It would also establish proof of principle that pre-treatment with oral prednisone is equally as efficacious as IV methylprednisolone.

The primary endpoint will be to assess the safety and tolerability of rituximab (Rituxan) in RA.

By showing that there are no differences in the frequency or severity of acute infusion reactions after rituximab when using pre-treatment with oral prednisone compared to I.V. methylprednisolone, we will establish proof of principle that oral prednisone is a viable alternative to I.V. methylprednisolone. Pre-treatment with oral prednisone would be a practical advantage for both the patient and the treating physician. The patient could self-administer this treatment at home thereby decreasing the time they would need to spend at the infusion center. Further, this dose of prednisone has fewer side effects than 100mg of methylprednisolone.

DETAILED DESCRIPTION:
This study will be an open-label prospective analysis of oral prednisone (compared to IV methylprednisolone) as a pre-treatment for rituximab in patients with rheumatoid arthritis. The study will be useful as pilot data to establish that there are no different trends between the two treatment strategies at decreasing the frequency and severity of acute infusion reactions. It would also establish proof of principle that pre-treatment with oral prednisone is equally as efficacious as IV methylprednisolone.

The primary endpoint will be to assess the safety and tolerability of rituximab (Rituxan) in RA.

By showing that there are no differences in the frequency or severity of acute infusion reactions after rituximab when using pre-treatment with oral prednisone compared to I.V. methylprednisolone, we will establish proof of principle that oral prednisone is a viable alternative to I.V. methylprednisolone. Pre-treatment with oral prednisone would be a practical advantage for both the patient and the treating physician. The patient could self-administer this treatment at home thereby decreasing the time they would need to spend at the infusion center. Further, this dose of prednisone has fewer side effects than 100mg of methylprednisolone..

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology Criteria for Rheumatoid Arthritis
* Age 18-80
* Concomitant methotrexate (MTX) [oral or parenteral at any dose]
* IgG & IgM levels above lower limit of normal.
* Adequate renal function as indicated by serum creatinine of < or = 1.8
* Study subjects can be either MTX-inadequate responders or TNF-alpha antagonists inadequate responders
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.
* If patients are on corticosteroids, they must be on a dose of < or = to prednisone 10mg oral daily (or its equivalence) and the dose must remain stable for 4 weeks prior to their first rituximab infusion.

Exclusion Criteria:

* An inflammatory arthritis other than RA
* ANC < 1.5 x 103
* Hemoglobin: < 8.0 gm/dL
* Platelets: < 100,000/mm
* AST or ALT >2.5 x Upper Limit of Normal unless related to primary disease.
* Positive Hepatitis B or C serology (Hep B Surface antigen and Hep C antibody)
* History of positive HIV (HIV conducted during screening if applicable)
* Treatment with any TNF-alpha antagonist within 8 weeks of Day 1 visit (for infliximab and adalimumab) or 4 weeks (for etanercept).
* Previous treatment with abatacept (Orencia) at any time.
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera® / Rituxan®)
* Previous treatment with Natalizumab (Tysabri®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Ongoing use of high dose steroids (>10mg/day) or unstable steroid dose in the past 4 weeks
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or lactation
* Concomitant malignancies or previous malignancies within 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Inability to comply with study and follow-up procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Carter, M.D., Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - University of South Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2008 to January 2011 in the medical clinic.
Pre-assignment Details: All study participants were treated with open-label standard dose and the recommended infusions of rituximab for rheumatoid arthritis.
Groups:
- Oral Prednisone as a Pretreatment to Rituximab: 40mg of oral prednisone given 30 min prior to rituximab as a prophylaxis against acute infusion reactions(AIR), as an alternative to the intravenous methylprednisone as a pretreatment for rituximab.
Period: Overall Study
Arm/Group | Oral Prednisone as a Pretreatment to Rituximab
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral Prednisone as a Pretreatment to Rituximab
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Acute Infusion Reactions in the First 24 Hours After Oral Prednisone Pretreatment to Initial Rituximab Infusion
Description: Open-label assessment of AIR's during and/or within 24 hours in patients pretreated with 40mg oral prednisone 30 minutes prior to initial rituximab infusion
Time Frame: 24 hours
Population: The subjects were 18-80 years of age, and fulfilled the 1987 American College of Rheumatology Criteria for Rheumatoid Arthritis, and taking concomitant methotrexate.
Measure: Number; unit: acute infusion reactions
Arm/Group | Oral Prednisone as a Pretreatment to Rituximab
Number analyzed (Participants) | 50
acute infusion reactions | 50

2. Secondary Outcome: Adverse Infusion Reactions Within 24 Hours Following the Second Rituximab Infusion.
Description: Assessment of all adverse infusion reactions within 24 hours of receipt of the second rituximab infusion
Time Frame: 24 hours
Measure: Number; unit: acute infusion reactions
Arm/Group | Oral Prednisone as a Pretreatment to Rituximab
Number analyzed (Participants) | 48
acute infusion reactions | 48

3. Secondary Outcome: Adverse Events Assessed From Day 15 Through Week 26.
Description: All adverse events reported from day 15 (24 hours after second infusion) through week 26.
Time Frame: 24 weeks
Measure: Number; unit: events
Arm/Group | Oral Prednisone as a Pretreatment to Rituximab
Number analyzed (Participants) | 48
events | 48

ADVERSE EVENTS:
Arm/Group | Oral Prednisone as a Pretreatment to Rituximab
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 32/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Prednisone as a Pretreatment to Rituximab (N=50)
atrial fibrillation (Cardiac disorders) | 1 (1)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (50)
suicide attempt (Psychiatric disorders) | 1 (50)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Prednisone as a Pretreatment to Rituximab (N=50)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 12
sinusitis (Respiratory, thoracic and mediastinal disorders) | 3
headache (General disorders) | 3
backache (Musculoskeletal and connective tissue disorders) | 2
diarrhea (Gastrointestinal disorders) | 2
fall (Injury, poisoning and procedural complications) | 2
fibromyalgia flare (Nervous system disorders) | 2
fracture (Musculoskeletal and connective tissue disorders) | 2
nausea (Gastrointestinal disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
An area of weakness to the study was the lack of direct comparison group.This was a single university study with two sites the cost,practicality of performing a noninferiority trial comparing these two pretreatment strategies was not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less